CLINICAL TRIAL: NCT06640868
Title: Pilot Sequential Multiple Assignment Randomized Trial for RSV Vaccine Uptake in Pregnancy
Brief Title: Promotion of RSV Immunization Through Multiple Efforts
Acronym: PRIME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jeannie Kelly, Associate Professor, Washington University School of Medicine
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 202408045
Record Dates: First submitted 2024-09-30; First posted 2024-10-15 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy; Vaccination
Keywords: RSV vaccine in pregnancy; vaccine uptake in pregnancy; sequential multiple assignment randomized trial
MeSH Terms: interventions — Audiovisual Aids

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Routine counseling (No Intervention): Randomized to routine counseling at 28-30 weeks
- Routine counseling + MyChart nurse managing (Active Comparator): Randomized to routine counseling at 28-30 weeks; not vaccinated by 34 weeks, and randomized to receive a MyChart message from the nurse encouraging vaccination at 34 weeks
  Interventions: Behavioral: MyChart nurse message
- Routine counseling + SMFM video (Active Comparator): Randomized to routine counseling at 28-30 weeks; not vaccinated by 34 weeks, and randomized to watch the SMFM video on RSV vaccination at a prenatal visit at 34 weeks
  Interventions: Behavioral: SMFM video
- Routine counseling/visual aid (Active Comparator): Randomized to routine counseling and receipt of a visual aid encouraging RSV vaccination at 28-30 weeks
  Interventions: Behavioral: Visual aid
- Routine counseling/visual aid + MyChart nurse message (Active Comparator): Randomized to routine counseling and receipt of a visual aid encouraging RSV vaccination at 28-30 weeks; not vaccinated by 34 weeks, and randomized to receive a MyChart message from the nurse encouraging vaccination at 34 weeks
  Interventions: Behavioral: MyChart nurse message; Behavioral: Visual aid
- Routine counseling/visual aid + SMFM video (Active Comparator): Randomized to routine counseling and receipt of a visual aid encouraging RSV vaccination at 28-30 weeks; not vaccinated by 34 weeks, and randomized to watch the SMFM video on RSV vaccination at a prenatal visit at 34 weeks
  Interventions: Behavioral: SMFM video; Behavioral: Visual aid

INTERVENTIONS:
Behavioral: MyChart nurse message — Receipt of a MyChart nurse message around 34 weeks encouraging RSV vaccination
  Arms: Routine counseling + MyChart nurse managing; Routine counseling/visual aid + MyChart nurse message
Behavioral: SMFM video — Receipt of SMFM video around 34 weeks encouraging RSV vaccination
  Arms: Routine counseling + SMFM video; Routine counseling/visual aid + SMFM video
Behavioral: Visual aid — Receipt of a visual aide encouraging RSV vaccination at 28-30 wks
  Arms: Routine counseling/visual aid; Routine counseling/visual aid + MyChart nurse message; Routine counseling/visual aid + SMFM video

SUMMARY:
Central hypothesis: a multimodal approach is needed to enhance RSV vaccine uptake in pregnancy rather than the current standard of care that relies solely on physician recommendations at routine prenatal visits and/or mass messaging to the public. The investigators propose a pilot sequential multiple assignment randomized trial (SMART) to evaluate the effectiveness of a bundle of evidence-based and sequential strategies to test early (28-30 weeks gestation) and late (34-36 weeks gestation efficacy) to increase RSV vaccination during pregnancy.

DETAILED DESCRIPTION:
Respiratory syncytial virus (RSV) is the leading cause of hospitalization and death among infants. Each year, up to 80,000 children are hospitalized due to RSV-associated lower respiratory tract infection, with infants having the highest risk. 50% of childhood deaths from RSV are in infants <6 months old. 1 in every 28 deaths among children aged 28 days to 6 months are attributed to RSV. Childhood RSV is also associated with long-term morbidity particularly a 12-fold higher risk of developing asthma. RSV prevention strategies are urgently needed to protect young infants particularly given their vulnerable immunity at birth. Passive immunity via transfer of IgG antibodies from immunized pregnant women offers an evidence-based solution and is endorsed by the American College of Obstetricians and Gynecologists and the Centers for Disease Control. In 2023, the FDA approved the RSVpreF vaccine for use during 32-36 weeks of pregnancy to protect infants from RSV-associated respiratory infection.

Despite the availability of the RSVpreF vaccine and formal guidelines recommending this vaccine in pregnancy during the 2023 RSV season, RSV vaccine uptake among pregnant individuals at our center was astoundingly low. In a review of 676 eligible patients, less than 10% received the RSV vaccine. Similar trends were seen with the COVID-19 and influenza vaccines in pregnancy where pregnant individuals were vaccinated at half of the rate of non-pregnant individuals. General barriers and facilitators for antenatal vaccine uptake have been well studied and are centered on provider recommendation, women's knowledge and beliefs about the safety of the vaccine, and logistical barriers such as on site availability. However, a recent initiative to offer on-site COVID-19 vaccination at a high risk pregnancy clinic resulted in only a 3% uptake of the vaccine among eligible, high-risk obstetric patients, suggesting that vaccine hesitancy, not availability, is a critical driver of the low vaccination rates in this population. Therefore, novel and multiple interventions are needed to address patient motivation and hesitancy, in addition to vaccine availability, to optimize vaccine uptake in pregnancy.

The central hypothesis is that a multimodal approach is needed to enhance RSVpreF vaccine uptake in pregnancy rather than the current standard of care that relies solely on physician recommendations at routine prenatal visits and/or mass messaging to the public. The investigators propose a pilot sequential multiple assignment randomized trial (SMART) to evaluate the effectiveness of a bundle of evidence-based and sequential strategies and test the following aims:

Aim 1: Assess the effectiveness of early (28-30 week) and low-intensity interventions to increase prenatal RSV vaccination uptake The investigators will compare vaccination uptake rates among pregnant patients 28-30 weeks gestation who are randomized to receive one of two low-intensity and universally acceptable interventions: physician counseling at prenatal visits vs routine counseling + patient visual aid administration (Figure 1). The investigators hypothesize that the combination of a visual aid with routine counseling will increase vaccination uptake rates by 34 weeks gestation. The investigators will explore whether demographic, clinical, or psychosocial factors modify the effects of each intervention.

Aim 2: Assess the effectiveness of late (34-36 week) higher-intensity interventions to increase prenatal RSV vaccination uptake for those who remain unvaccinated at 34 weeks gestation. The investigators will compare vaccination uptake rates in patients who remain unvaccinated at 34 weeks between two higher-intensity interventions: targeted patient phone calls encouraging vaccination versus individual physician reminders on the day of patient appointment. The investigators hypothesize that targeted patient calls will result in the highest vaccination uptake rates due to prior literature supporting the efficacy of this intervention. The investigators will explore whether demographic, clinical, or psychosocial factors modify the effects of each intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed intrauterine pregnancy (IUP) at 28-30 weeks.
2. No contraindications to the RSV vaccine: history of severe allergic reaction to any vaccine component or active moderate/severe acute illness with or without fever or receipt of RSV vaccine during the pregnancy

Exclusion Criteria:

* Those who do not have confirmed IUP at 28-30 weeks, or who have a contraindication to the RSV vaccine (history of severe allergic reaction to any vaccine component or active moderate/severe acute illness with or without fever or receipt of RSV vaccine during the pregnancy) will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Vaccinated for RSV by delivery | Between 32 weeks and delivery, usually around 40 weeks gestation
  Vaccinated for RSV by delivery
Feasibility Outcomes | From time of randomization through delivery; at most will be 15 weeks
  Percent of patients eligible for Tier 1 randomization receiving randomization; Percent of patients eligible for Tier 2 randomization receiving randomization; Number of patients delivered prior to Tier 2 randomization, Number of patients assigned in Tier 1 and Tier 2 randomization receiving assignment, Number of patients declining assignment, Timeline for completion of N=50

SECONDARY OUTCOMES:
Vaccinated for RSV by 34 weeks | Pregnancy by 34 weeks
  Vaccinated for RSV by 34 weeks
Receipt of Tdap during pregnancy | Between 27 weeks and delivery, usually around 40 weeks gestation
  Receipt of Tdap during pregnancy
Receipt of Flu vaccine during pregnancy | During pregnancy, usually 40 weeks long
  Receipt of Flu vaccine during pregnancy
Receipt of COVID vaccine during pregnancy | During pregnancy, usually 40 weeks long
  Receipt of COVID vaccine during pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No